CLINICAL TRIAL: NCT03036254
Title: Hyperbaric Oxygen Therapy for Cognition in Diabetic Elderly at High Dementia Risk
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Icahn School of Medicine at Mount Sinai (Other)
Collaborators: Sheba Medical Center (Other Government); Assaf-Harofeh Medical Center (Other Government); University of Wisconsin, Madison (Other)
Responsible Party: Principal Investigator, Michal Beeri, Professor, Psychiatry, Icahn School of Medicine at Mount Sinai
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: GCO 15-0192
Record Dates: First submitted 2017-01-25; First posted 2017-01-30 (Estimated); Results first posted 2025-08-11 (Actual); Last update posted 2025-08-11 (Actual); Status verified 2025-07

CONDITIONS: Diabetes Mellitus
Keywords: Diabetes Mellitus; Cognition
MeSH Terms: conditions — Diabetes Mellitus | interventions — Hyperbaric Oxygenation

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- HBOT intervention (Experimental): The multiplace HBOT unit at Asaf Harofeh. The inside looks like an airplane, with comfortable chairs for 11 subjects and the nurse who stays throughout the session. The HBOT protocol is 90 minutes, 5 times/week, 60 sessions, 100% oxygen at 2 ATA with 5 minute air breaks every 30 minutes.
  Interventions: Device: HBOT intervention
- Sham intervention (Sham Comparator): Except for pressure, all the conditions of the HBOT intervention are provided in the sham intervention (nurse measures vitals and asks about health before entering the chamber, time in the chamber, number of sessions per week and overall, nurse in the chamber at all times, mask on the face, etc.).
  Interventions: Device: HBOT intervention; Device: Sham intervention

INTERVENTIONS:
Device: HBOT intervention — HBOT is a treatment in which oxygen-enriched air (up to 100%) is administered to patients at a pressure.
  HBOT intervention arm - 3 months of HBOT treatment, 9 months observation
  all participants receive HBOT treatment for 3 months at year 2
  Other Names: Hyperbaric oxygen therapy
Device: Sham intervention — Sham was selected as the control condition rather than "usual care" to equate intervention groups with respect to other variables that could influence cognition and functional status, such as a new challenge (completing an activity program), peer socialization, and attention from staff.
  Arms: Sham intervention

SUMMARY:
An urgent need exists to identify effective interventions to arrest or reverse dementia and cognitive loss at its earliest stages. The proposed pilot randomized clinical trial will investigate the short and long-term effects of hyperbaric oxygen therapy on cognitive functioning, cerebral blood flow, and glucose uptake in diabetic elderly with mild cognitive impairment. and provide the basis for a large-scale multi-center study of hyperbaric oxygen therapy effects on cognition in diabetes. The potential to preserve, or even enhance, cognition in elderly at high risk of cognitive decline and dementia has major implications for the affected individuals and their support systems that bear the social and financial burdens of long-term caregiving.

DETAILED DESCRIPTION:
This resubmission responds to "PAR-16-365-Pilot Clinical Trials for the Spectrum of Alzheimer's Disease and Age-related Cognitive Decline (R01)". It will examine the efficacy of hyperbaric oxygen therapy (HBOT) in improving cognitive functioning in cognitively impaired elderly with diabetes (T2D), who have high risk for dementia. It is a collaboration of the Icahn School of Medicine at Mount Sinai, NY, the University of Wisconsin, the Sagol Center for Hyperbaric Medicine and Research at Asaf Harofeh Medical Center, Israel-one of the world's largest and busiest hyperbaric units-and the Sheba Medical Center, Israel.

HBOT is a treatment in which oxygen-enriched air (up to 100%) is administered to patients at a pressure above the ambient atmosphere. The combined action of hyperoxia and hyperbaric pressure leads to significant improvements in tissue oxygenation, resulting in cerebrovascular benefits with improved ischemic damage and cerebral blood flow. Recently, the researchers of this group published compelling evidence from clinical trials indicating HBOT neurotherapeutic effects in stroke, with better cognitive function and elevated brain activity in SPECT. New preliminary data suggests potential neurotherapeutic effects of HBOT on T2D elderly with mild cognitive impairment (MCI), showing better cognitive performance and brain activity. The researchers propose a randomized controlled clinical trial examining the short (12 weeks) and long-term (12 months) efficacy of HBOT. The researchers will test hypotheses that HBOT compared to a sham condition improves cognitive function and increases cerebral blood flow and glucose utilization in MCI patients with T2D. Such patients are at high dementia risk and enriched in cerebrovascular disease, and thus have high potential for benefitting from HBOT. Aim 1 examines the potential beneficial effects of HBOT on cognition (with a primary composite measure of executive functions and episodic memory, both affected by T2D). Aim 2 examines effects of HBOT on ischemic injury which will be measured by CBF at the level of capillaries in gray matter (by MRI arterial spin labeling), and in macrovessels (by a novel 4D Flow MRI technology developed by the researchers of this group). Aim 3 focuses on effects of HBOT on cerebral glucose utilization using [F18]FDG-PET. Finally, Aim 4 investigates mediation by the biomarkers, i.e. whether their inclusion in a mediation model will attenuate the effect of HBOT on cognition, suggesting them as underlying mechanisms. This study will be performed in Israel, where there is optimal infrastructure and expertise for all the study components at significantly lower costs. HBOT can be widely deployed in the US so if successful, this pilot study will provide the basis for a multi-center large-scale clinical trial for definitive evidence of its benefits to cognition in T2D patients at high dementia risk. Despite advances in the understanding of risk factors and the pathologic basis for dementia, treatments are of very limited effects. As the proportion of elderly increases, the accelerating prevalence of T2D and dementia amplifies this application's public health impact.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of T2D
* Diagnosis of MCI
* > the age of 65
* Hebrew fluency
* An informant

Exclusion Criteria:

* Brain disease that affects cognition (e.g. Parkinson's disease, schizophrenia).
* Stroke
* Epilepsy
* Chest pathology incompatible with HBOT
* Inner ear disease
* Claustrophobia
* Cholinesterase inhibitors
* Subjects with an indication for HBOT
* Counter-indication for MRI or PET
* Individuals with severe cataracts must have cataract operations before enrolling in the study

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 155 (Actual)
Dates: Start 2017-08-10 (Actual); Primary Completion 2024-04-15 (Actual); Study Completion 2024-04-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michal Schnaider-Beeri, PhD, Principal Investigator — Icahn School of Medicine at Mount Sinai; Mary Sano, PhD, Principal Investigator — Icahn School of Medicine at Mount Sinai
Locations (4):
- United States (2):
  - Icahn School of Medicine at Mount Sinai, New York, New York
  - University of Wisconsin, Madison, Wisconsin
- Israel (2):
  - Sheba Medical Center, Ramat Gan
  - Assaf HaRofeh Medical Center, Tzrifin

IPD SHARING:
Plan to Share IPD: Yes
De-identified MRI and PET scans and cognitive scores will be made available for investigative collaborations. We expect to share these data with a large number of investigators throughout the world.

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 155 participants were enrolled from August 10, 2017, to April 17, 2023. The Covid-19 pandemic caused a 14-month pause, affecting follow-up numbers, but the trial was concluded successfully.
Groups:
- HBOT Intervention: The multiplace HBOT unit at Asaf Harofeh. The inside looks like an airplane, with comfortable chairs for 11 subjects and the nurse who stays throughout the session. The HBOT protocol is 90 minutes, 5 times/week, 60 sessions, 100% oxygen at 2 ATA with 5 minute air breaks every 20 minutes.
- Sham Intervention: The sham condition replicates all experiential aspects of the HBOT therapy except for the degree of pressure and oxygen levels. The sham condition exposes subjects to 1.1 ATA, which provides a pressure sensation in addition to the noise of air circulation. Pressure then decreases very slowly during the next half hour; in the last 5 minutes of the session, air is circulated again with its related noise.
Period: Overall Study
Arm/Group | HBOT Intervention | Sham Intervention
Started | 77 | 78
Completed | 60 | 67
Not Completed | 17 | 11
Not completed — Adverse Event | 6 | 4
Not completed — Death | 3 | 1
Not completed — Lack of Efficacy | 5 | 1
Not completed — Withdrawal by Subject | 3 | 5

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | HBOT Intervention | Sham Intervention | Total
Number analyzed (Participants) | 77 | 78 | 155
Age, Continuous [Mean (Standard Deviation); unit: years] | 71.7 (4.182) | 70.2 (3.560) | 70.94 (3.938)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 27 | 21 | 48
  Male | 50 | 57 | 107
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  MENA: Middle Eastern North African | 33 | 44 | 77
  Ashkenazi | 41 | 32 | 73
  Unknown | 3 | 2 | 5
Clinical Dementia Rating - Sum of Boxes (CDR-SB) [Mean (Standard Deviation); unit: units on a scale] — Total scale from 0-18. Higher score suggests more severe dementia.
  units on a scale | 1.6 (1.16) | 1.51 (0.80) | 1.56 (0.99)
Total Mini-Mental State Examination [Mean (Standard Deviation); unit: units on a scale] — Total scale from 0-30, with scores > 25 interpreted as normal cognitive status.
  units on a scale | 28.55 (1.28) | 28.49 (1.36) | 28.52 (1.32)
Total Beck Depression Inventory [Mean (Standard Deviation); unit: units on a scale] — Total score from 0-63. Higher score indicates more severe depressive symptoms.
  units on a scale | 5.52 (3.89) | 5.34 (4.02) | 5.43 (3.95)

OUTCOME MEASURES:

1. Primary Outcome: Change in Global Cognition Score
Description: This analysis involves 11 cognitive performance variables, each measuring a specific aspect of cognition. In general, higher scores indicate better performance (Digit Symbol measures processing speed, Semantic Fluency measures verbal fluency, Word Recall Task measures immediate verbal memory, Delayed Word Recall Test measures delayed verbal memory, and Recall Unit measures immediate and delayed story recall), except for two variables (Trail Making Test Part A measures processing speed, Trail Making Test Part B measures cognitive flexibility) that measure time (where higher values indicate worse performance). These variables are standardized using Z-scores, which allow for combining and comparing values across different scales.
  The standardized values (Z-scores) of all 11 measures are averaged to create the composite score. Full range of composite score is -1 to 1. Higher composite Z-score reflects better cognitive performance and more favorable outcomes.
Time Frame: baseline, 12, weeks, 6 months and 12 months
Population: The Covid-19 pandemic caused a 14-month pause, affecting follow-up numbers.
Measure: Mean (Standard Deviation); unit: Composite z-score
Arm/Group | HBOT Intervention | Sham Intervention
Number analyzed (Participants) | 77 | 78
Composite z-score
  Visit 1 - Baseline: number analyzed (Participants) | 76 | 78
  Visit 1 - Baseline | -0.012 (0.65) | 0.021 (0.61)
  Visit 2 - 12 weeks: number analyzed (Participants) | 64 | 62
  Visit 2 - 12 weeks | 0.18 (0.67) | 0.32 (0.73)
  Visit 3 - 6 months: number analyzed (Participants) | 57 | 54
  Visit 3 - 6 months | 0.38 (0.68) | 0.48 (0.64)
  Visit 4- 12 months: number analyzed (Participants) | 64 | 65
  Visit 4- 12 months | 0.34 (0.65) | 0.37 (0.77)

2. Primary Outcome: Cerebral Blood Flow
Description: Cerebral blood flow (CBF) via arterial spin labeling magnetic resonance imaging (ASL-MRI). CBF is defined as the blood volume that flows per unit mass per unit time in brain tissue.
Time Frame: baseline, 3 months, and 12 months
Population: The Covid-19 pandemic caused a 14-month pause, affecting follow-up numbers
Measure: Mean (Standard Deviation); unit: ml blood∕100 g tissue min
Arm/Group | HBOT Intervention | Sham Intervention
Number analyzed (Participants) | 77 | 78
ml blood∕100 g tissue min
  Baseline: number analyzed (Participants) | 48 | 47
  Baseline | 219.39 (60.92) | 207.86 (83.50)
  3 months: number analyzed (Participants) | 41 | 42
  3 months | 227.68 (68.67) | 227.64 (49.02)
  12 months: number analyzed (Participants) | 51 | 51
  12 months | 216.91 (50.54) | 216.91 (50.54)

3. Primary Outcome: Whole Brain SUVr (FDG-PET)
Description: Measures how actively the brain uses glucose, highlighting areas with abnormal activity that may signal diseases like Alzheimer's. Dimmer areas suggest reduced activity seen in disorders like dementia.
Time Frame: Baseline, 12 weeks, 12 months
Population: The Covid-19 pandemic caused a 14-month pause, affecting follow-up numbers
Measure: Mean (Standard Deviation); unit: Standardized Uptake Value (SUV)
Arm/Group | HBOT Intervention | Sham Intervention
Number analyzed (Participants) | 77 | 78
Standardized Uptake Value (SUV)
  Visit 1 - Baseline: number analyzed (Participants) | 48 | 42
  Visit 1 - Baseline | 0.009 (0.907) | -0.022 (1.117)
  Visit 2 - 12 weeks: number analyzed (Participants) | 29 | 27
  Visit 2 - 12 weeks | -0.128 (1.265) | 0.379 (0.973)
  Visit 4 - 12 months: number analyzed (Participants) | 11 | 16
  Visit 4 - 12 months | -0.266 (0.934) | -0.0004 (0.828)

4. Secondary Outcome: NIH Computerized Cognitive Test
Description: The sum z-scores for 3 computer-based tests (not language dependent), developed through NIH; EXAMINER assessing executive abilities: http://examiner.ucsf.edu).
  Early in the study, it became clear that participants-older adults with significant frailty, multiple chronic conditions (average >4 per participant), and high medication burden (mean >5 medications)-were finding the assessment protocol burdensome.
  The protocol already required repeated cognitive testing, MRI, FDG-PET imaging, and other assessments, leading many participants to report fatigue and difficulty concentrating. To prioritize participant well-being, decision made not to add the NIH computerized cognitive tests. The existing paper-and-pencil battery was well-established, sensitive to cognitive changes, and adequately covered executive function and episodic memory.
  The NIH computerized cognitive test was never administered, and no data was collected at any time.
Time Frame: Baseline, 12 weeks, 6 months, 12 months
Population: Data not collected due to decision not to administered instruments. This decision was based on participant frailty and protocol intensity-not technical issues or non-compliance-and was made to ensure feasibility and ethical conduct of the study.
  The NIH computerized cognitive test was never administered, and no data was collected at any time.
Arm/Group | HBOT Intervention | Sham Intervention
Number analyzed (Participants) | 0 | 0

5. Secondary Outcome: Clinical Dementia Rating-Sum of Boxes (CDR-SB)
Description: Clinical Dementia Rating-Sum of Boxes (CDR-SB), which summarizes impairment in 6 domains (memory, orientation, judgment/problem solving, community affairs, home/hobbies, and personal care) based on subject and informant interviews. Scores in each of these are combined to obtain a composite score ranging from 0 (no symptoms of dementia) through 3 (severe symptoms of dementia).
  Total scale from 0-18. Higher scores indicating worse cognitive status.
Time Frame: baseline, 12, weeks, 6 months and 12 months
Population: The Covid-19 pandemic caused a 14-month pause, affecting follow-up numbers
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | HBOT Intervention | Sham Intervention
Number analyzed (Participants) | 77 | 78
score on a scale
  Baseline: number analyzed (Participants) | 75 | 78
  Baseline | 1.60 (1.16) | 1.51 (0.80)
  12 weeks: number analyzed (Participants) | 58 | 53
  12 weeks | 0.75 (0.86) | 0.67 (0.81)
  6 months: number analyzed (Participants) | 52 | 49
  6 months | 0.61 (0.62) | 0.76 (0.79)
  12 months: number analyzed (Participants) | 64 | 61
  12 months | 0.71 (0.75) | 0.87 (1.39)

6. Secondary Outcome: Beck Depression Inventory (BDI)
Description: This is a 21-item, self-report questionnaire that measures attitudes and symptoms of depression during the last week (i.e. mood, feelings of hopelessness, failure, guilt, self-esteem, etc.). Each question has a set of at least four possible responses, ranging in intensity. Total scale 0-63. Higher scores indicate more severe symptoms of depression.
Time Frame: baseline, 12 weeks, 6 months and 12 months
Population: The Covid-19 pandemic caused a 14-month pause, affecting follow-up numbers
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | HBOT Intervention | Sham Intervention
Number analyzed (Participants) | 77 | 78
score on a scale
  Baseline: number analyzed (Participants) | 75 | 78
  Baseline | 5.43 (3.8) | 5.31 (4.0)
  12 weeks: number analyzed (Participants) | 58 | 53
  12 weeks | 5.57 (4.80) | 4.74 (4.32)
  6 months: number analyzed (Participants) | 52 | 49
  6 months | 6.62 (6.51) | 4.88 (3.61)
  12 months: number analyzed (Participants) | 64 | 61
  12 months | 6.14 (5.8) | 5.64 (5.3)

7. Secondary Outcome: Alzheimer's Disease Cooperative Study-Activities of Daily Living - Prevention Questionnaire (ADL-PI)
Description: ADL questionnaire Participant
  The ADL-PI was developed, comprising 15 ADL (e.g. managing medications, managing finances) and 5 physical function (e.g. shopping and meal preparation) questions. All responses relate to the 3 months prior to the time of rating.
  Total range 0-30, higher scores indicate greater impairment.
Time Frame: baseline, 12 weeks, 6 months, and 12 months
Population: The Covid-19 pandemic caused a 14-month pause, affecting follow-up numbers
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | HBOT Intervention | Sham Intervention
Number analyzed (Participants) | 77 | 78
score on a scale
  Baseline: number analyzed (Participants) | 75 | 78
  Baseline | 24.34 (4.041) | 24.60 (3.81)
  12 weeks: number analyzed (Participants) | 58 | 53
  12 weeks | 25.43 (4.53) | 25.58 (3.99)
  6 months: number analyzed (Participants) | 52 | 49
  6 months | 25.71 (3.76) | 25.84 (4.00)
  12 months: number analyzed (Participants) | 64 | 61
  12 months | 26.29 (3.20) | 25.47 (4.02)

8. Secondary Outcome: Alzheimer's Disease Cooperative Study-Activities of Daily Living - Mild Cognitive Impairment (ADCS-ADL MCI)
Description: ADL Informant
  This tool is based on caregiver's report to assess participants' abilities to perform basic and instrumental activities of daily living (ADLs) like bathing, walking and self-grooming. All responses should relate to the 4 weeks prior to the time of rating. Full Scale range from 0-53, higher score indicates more impairment for the participant.
Time Frame: Baseline, 12 weeks, 6 months, and 12 months
Population: The Covid-19 pandemic caused a 14-month pause, affecting follow-up numbers
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | HBOT Intervention | Sham Intervention
Number analyzed (Participants) | 77 | 78
score on a scale
  Baseline: number analyzed (Participants) | 75 | 78
  Baseline | 45.24 (6.12) | 44.71 (5.9)
  12 weeks: number analyzed (Participants) | 58 | 53
  12 weeks | 47.5 (5.67) | 48.41 (4.49)
  6 months: number analyzed (Participants) | 52 | 49
  6 months | 47.69 (5.66) | 47.29 (5.33)
  12 months: number analyzed (Participants) | 64 | 61
  12 months | 48.98 (3.67) | 48.32 (6.07)

9. Secondary Outcome: Total Mini-Mental State Examination (MMSE)
Description: Total range 0-30, higher scores indicate better cognitive function.
Time Frame: Baseline, 12 weeks, 6 months, and 12 months
Population: The Covid-19 pandemic caused a 14-month pause, affecting follow-up numbers
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | HBOT Intervention | Sham Intervention
Number analyzed (Participants) | 77 | 78
score on a scale
  Baseline: number analyzed (Participants) | 75 | 78
  Baseline | 28.56 (1.30) | 28.49 (1.37)
  12 weeks: number analyzed (Participants) | 58 | 53
  12 weeks | 28.26 (1.63) | 28.38 (1.77)
  6 months: number analyzed (Participants) | 52 | 49
  6 months | 28.04 (1.89) | 28.53 (1.53)
  12 months: number analyzed (Participants) | 64 | 61
  12 months | 28.32 (1.68) | 28.18 (2.21)

ADVERSE EVENTS:
Time Frame: 12 months
Arm/Group | HBOT Intervention | Sham Intervention
All-Cause Mortality (participants affected / at risk) | 3/77 | 1/78
Serious Adverse Events (participants affected / at risk) | 18/77 | 6/78
Other Adverse Events (participants affected / at risk) | 55/77 | 51/78
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | HBOT Intervention (N=77) | Sham Intervention (N=78)
Acute cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Barotrauma (Injury, poisoning and procedural complications) | 1 | 0
Bypass surgery (Surgical and medical procedures) | 1 | 0
Cardiac Arrythmia (Cardiac disorders) | 0 | 1
Cardiac catheterization (Surgical and medical procedures) | 3 | 0
Chest pain (General disorders) | 1 | 0
Deceased (General disorders) | 3 | 1
Dizziness (Nervous system disorders) | 0 | 1
Fall (Injury, poisoning and procedural complications) | 1 | 1
Inguinal hernia (Gastrointestinal disorders) | 1 | 1
Intracranial pressure increase (Nervous system disorders) | 1 | 0
Knee arthroplasty (Surgical and medical procedures) | 1 | 0
Lung cancer stage IV (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Metatarsal fracture (Injury, poisoning and procedural complications) | 1 | 0
Myocardial infarction (Cardiac disorders) | 1 | 1
Parathyroidectomy (Surgical and medical procedures) | 1 | 0
Pneumonia (Infections and infestations) | 1 | 1
Retinal detachment (Eye disorders) | 2 | 0
Shoulder replacement (Surgical and medical procedures) | 1 | 0
Stroke (Nervous system disorders) | 2 | 1
Syncope (Nervous system disorders) | 1 | 0
Urinary infection (Infections and infestations) | 1 | 0
Weakness (General disorders) | 0 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | HBOT Intervention (N=77) | Sham Intervention (N=78)
Abscess in the throat (Infections and infestations) | 0 | 1
Acoustic neuromas (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Ankle fracture (Injury, poisoning and procedural complications) | 0 | 1
Arachnoid granulation (Nervous system disorders) | 0 | 1
Atrial fibrilation (Cardiac disorders) | 0 | 2
Atrial fibrillation (Cardiac disorders) | 0 | 2
Avastin eye injection (Eye disorders) | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 5 | 1
Bacteremia (Infections and infestations) | 1 | 0
Barotrauma (Injury, poisoning and procedural complications) | 20 | 4
Basalioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
BDI=22 (Psychiatric disorders) | 0 | 1
Blurry vision (Eye disorders) | 0 | 1
Bone spur (Musculoskeletal and connective tissue disorders) | 0 | 1
Bronchitis (Infections and infestations) | 2 | 0
Bruised ear (Injury, poisoning and procedural complications) | 1 | 0
Cardiac catheterization (Surgical and medical procedures) | 3 | 1
Cataract (Eye disorders) | 6 | 2
Cavernoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Chest pain (General disorders) | 2 | 0
Claustrophobia (Psychiatric disorders) | 1 | 0
Cold (Infections and infestations) | 2 | 2
Colon inflammation (Gastrointestinal disorders) | 1 | 0
Colonoscopy (Surgical and medical procedures) | 1 | 0
Conjunctivitis (Eye disorders) | 0 | 1
Covid 19 (Infections and infestations) | 10 | 9
Diabetic foot ulcer (Musculoskeletal and connective tissue disorders) | 0 | 1
Diplopia (Eye disorders) | 1 | 0
Dizziness (Nervous system disorders) | 0 | 1
Essential tremor (Nervous system disorders) | 0 | 1
Exacerbation of post traumatic symptoms (BDI=24) (Psychiatric disorders) | 1 | 0
Eye pain (Eye disorders) | 1 | 0
Facial paralysis (Nervous system disorders) | 1 | 0
Fall (Injury, poisoning and procedural complications) | 5 | 4
Fasciculation (Nervous system disorders) | 0 | 1
Fracture of the coccyx (Injury, poisoning and procedural complications) | 0 | 1
Glaucoma (Eye disorders) | 1 | 0
Gum infection (Infections and infestations) | 0 | 1
Hand tendon injury (Injury, poisoning and procedural complications) | 1 | 0
Head injury (Injury, poisoning and procedural complications) | 1 | 0
Herpes zoster (Infections and infestations) | 0 | 1
Hip injury (Injury, poisoning and procedural complications) | 1 | 2
Hip replacement (Surgical and medical procedures) | 0 | 1
Hyperglycemia (Metabolism and nutrition disorders) | 0 | 1
Hypertension (Vascular disorders) | 3 | 0
Hypothermia (General disorders) | 0 | 1
Inguinal hernia (Gastrointestinal disorders) | 0 | 4
Itchy skin (Skin and subcutaneous tissue disorders) | 1 | 0
Joint pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Kidney stones (Renal and urinary disorders) | 1 | 0
Knee effusion (Musculoskeletal and connective tissue disorders) | 1 | 0
Knee fracture (Injury, poisoning and procedural complications) | 0 | 1
Lumbar disc herniation (Musculoskeletal and connective tissue disorders) | 1 | 1
Lumbar puncture (Surgical and medical procedures) | 1 | 1
Metatarsal fracture (Injury, poisoning and procedural complications) | 0 | 1
MRI brain abnormal (Investigations) | 1 | 1
Myringotomy (Surgical and medical procedures) | 1 | 0
Nausea (Gastrointestinal disorders) | 0 | 1
Neuropathy (Nervous system disorders) | 1 | 0
Osteoporosis (Musculoskeletal and connective tissue disorders) | 0 | 1
Pains in legs (Musculoskeletal and connective tissue disorders) | 1 | 0
Parkinson's disease (Nervous system disorders) | 0 | 1
Pneumonia (Infections and infestations) | 0 | 1
Post traumatic pain (Injury, poisoning and procedural complications) | 0 | 1
Post-traumatic stress disorder (Psychiatric disorders) | 1 | 0
Posture abnormal (Musculoskeletal and connective tissue disorders) | 0 | 1
Prostate resection (Surgical and medical procedures) | 1 | 3
Pulmonary granuloma (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Shoulder fracture (Injury, poisoning and procedural complications) | 0 | 1
Shoulder replacement (Surgical and medical procedures) | 1 | 0
Sinusitis (Infections and infestations) | 0 | 2
Skin cyst (Skin and subcutaneous tissue disorders) | 2 | 0
Skin infection (Skin and subcutaneous tissue disorders) | 0 | 1
Sleep apnea (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Stomach ache (Gastrointestinal disorders) | 0 | 2
Stroke (Nervous system disorders) | 1 | 0
Syncope (Nervous system disorders) | 1 | 0
Tinnitus (Ear and labyrinth disorders) | 0 | 1
Trigger finger (Musculoskeletal and connective tissue disorders) | 0 | 1
Vertigo (Ear and labyrinth disorders) | 1 | 0
Vision decreased (Eye disorders) | 2 | 1
Vitreous detachment (Eye disorders) | 1 | 0
Vomiting (Gastrointestinal disorders) | 0 | 3
Weakness (General disorders) | 0 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
There is an agreement between the sponsor (or its agent) and any non-employee PI(s) that restricts the PI's rights to discuss or publish trial results after the Primary Completion Date.

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2020-05-21): https://cdn.clinicaltrials.gov/large-docs/54/NCT03036254/Prot_SAP_000.pdf
  • Informed Consent Form (2022-01-05): https://cdn.clinicaltrials.gov/large-docs/54/NCT03036254/ICF_001.pdf